CLINICAL TRIAL: NCT02325401
Title: A Phase I Dose-finding Study of Metformin in Combination With Concurrent Cisplatin and Radiation in Patients With Locally Advanced Head and Neck Squamous Cell Carcinoma
Brief Title: Dose-finding Study of Metformin With Chemoradiation in Locally Advanced Head and Neck Squamous Cell Carcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, Trisha Wise-Draper, Principal Investigator, University of Cincinnati
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCCI-HN-14-01
Record Dates: First submitted 2014-12-16; First posted 2014-12-25 (Estimated); Results first posted 2020-06-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-05

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Metformin; Cisplatin; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Metformin with Chemoradiation (Experimental): Metformin administered orally daily to start one week prior to Cisplatin and Radiation Therapy. Metformin dose is escalating.
  Interventions: Drug: Metformin; Drug: Cisplatin; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Metformin — Escalating doses of 2000mg, 2550 mg and 3000mg. Starting 1 week prior to the initiation of chemoradiation and ending the final day of chemo or radiation.
  Other Names: Fortamet; Glucophage; Glucophage XR; Glumetza; Riomet
Drug: Cisplatin — Dosed at 100mg/m2 on days 1, 22, and 43
  Other Names: Platinol; Platinol-AQ
Radiation: Radiation Therapy — 70 Gy in 2 Gy once daily fractions of 35 fractions

SUMMARY:
The purpose of this research study is to test the safety of adding metformin to standard of care. The standard of care treatment will be cisplatin once every 3 weeks for 3 treatments and radiation for 7 weeks.

Metformin is a medication that is currently used to treat diabetes. Increasing amounts of metformin will be given to groups of patients already receiving normal treatment for their cancer to see if metformin causes any good effects by killing your cancer or bad effects (side effects).

DETAILED DESCRIPTION:
Patients were registered by contacting the University of Cincinnati Clinical Trials Office. Patients must be registered and consent obtained prior to initiation of any protocol therapy.

Treatment was administered on an outpatient basis. Adverse events and potential risks for metformin and cisplatin and radiation were reported.

Patients must have screening labs performed within 2 weeks of start of treatment including a complete blood count, liver function tests, metabolic renal panel including magnesium, vitamin B12 level, lactate, and C-peptide. Renal panel must be verified within 24 hours of cisplatin administration. They must fulfill inclusion criteria.

The recommended starting dose of metformin in diabetic patients is 500mg orally twice a day which can be escalated by 500mg increments weekly as tolerated with the maximum recommended daily dose of 2550mg.

Cisplatin was given either before or after the radiation therapy fraction that is given on the same day. If radiation is held for more than 2 days (for any reason), cisplatin may be held as well until radiation resumes.

The prescribed radiotherapy dose was be 70 Gy in 2 Gy once-daily fraction size (total of 35 fractions).

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced squamous cell cancer of the head and neck, stage III or IV disease (T1-2, N2a-3 or T3-4).
* Measurable disease
* No prior chemotherapy or radiation for head and neck squamous cell cancer
* Life expectancy of greater than 3 months.
* Adequate labs

Exclusion Criteria:

* Known metastatic disease.
* Nasopharyngeal carcinoma
* History of allergic reactions attributed to metformin or other agents used in study.
* Known diagnosis of diabetes requiring insulin for control.
* Administration of metformin within last 4 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-05-11 (Actual); Primary Completion 2017-12-26 (Actual); Study Completion 2020-02-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Trisha Wise-Draper, MD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati Cancer Institute, Cincinnati, Ohio, United States

REFERENCES:
- [Derived] Crist M, Yaniv B, Palackdharry S, Lehn MA, Medvedovic M, Stone T, Gulati S, Karivedu V, Borchers M, Fuhrman B, Crago A, Curry J, Martinez-Outschoorn U, Takiar V, Wise-Draper TM. Metformin increases natural killer cell functions in head and neck squamous cell carcinoma through CXCL1 inhibition. J Immunother Cancer. 2022 Nov;10(11):e005632. doi: 10.1136/jitc-2022-005632. PMID 36328378

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were 18 years or old, with newly diagnosis LAHNSCC and ECOG rating of better than or equal to 1, with adequate organ function. Individuals were excluded if they had a diagnosis of: nasopharyngeal cancer, metastatic disease, diabetes requiring insulin, or receipt of metformin with in the last 4 weeks, or history of intercurrent illness.
Groups:
- Metformin (2000mg) With Chemoradiation: Metformin administered orally daily to start one week prior to Cisplatin and Radiation Therapy. Metformin dose is escalating. This is the 2000mg cohort.
- Metformin (2550mg) With Chemoradiation: Metformin administered orally daily to start one week prior to Cisplatin and Radiation Therapy. Metformin dose is escalating. This is the 2550mg cohort.
- Metformin (3000mg) With Chemoradiation: Metformin administered orally daily to start one week prior to Cisplatin and Radiation Therapy. Metformin dose is escalating. This is the 3000mg cohort.
Period: Overall Study
Arm/Group | Metformin (2000mg) With Chemoradiation | Metformin (2550mg) With Chemoradiation | Metformin (3000mg) With Chemoradiation
Started | 6 | 9 | 5
Completed | 6 | 8 | 4
Not Completed | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: There is a total of 18 participants in three cohorts: Metformin (2000mg) (n = 6); Metformin (2500mg) (n = 8); Metformin (3000mg) (n = 4).
Arm/Group | Metformin With Chemoradiation
Number analyzed (Participants) | 18
Age, Continuous [Median (Full Range); unit: Years] — Population: There is a total of 18 participants in three cohorts: Metformin (2000mg) (n = 6); Metformin (2500mg) (n = 8); Metformin (3000mg) (n = 4).
  Years
    Metformin (2000mg) With Chemoradiation: number analyzed (Participants) | 6
    Metformin (2000mg) With Chemoradiation | 54 [47 to 62]
    Metformin (2550mg) With Chemoradiation: number analyzed (Participants) | 8
    Metformin (2550mg) With Chemoradiation | 55.5 [46 to 65]
    Metformin (3000mg) With Chemoradiation: number analyzed (Participants) | 4
    Metformin (3000mg) With Chemoradiation | 53 [34 to 64]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: There is a total of 18 participants in three cohorts: Metformin (2000mg) (n = 6); Metformin (2500mg) (n = 8); Metformin (3000mg) (n = 4).
  Participants
    Metformin (2000mg) With Chemoradiation: number analyzed (Participants) | 6
    Metformin (2000mg) With Chemoradiation: Female | 1
    Metformin (2000mg) With Chemoradiation: Male | 5
    Metformin (2550mg) With Chemoradiation: number analyzed (Participants) | 8
    Metformin (2550mg) With Chemoradiation: Female | 0
    Metformin (2550mg) With Chemoradiation: Male | 8
    Metformin (3000mg) With Chemoradiation: number analyzed (Participants) | 4
    Metformin (3000mg) With Chemoradiation: Female | 2
    Metformin (3000mg) With Chemoradiation: Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: There is a total of 18 participants in three cohorts: Metformin (2000mg) (n = 6); Metformin (2500mg) (n = 8); Metformin (3000mg) (n = 4).
  Participants
    Metformin (2000mg) With Chemoradiation: number analyzed (Participants) | 6
    Metformin (2000mg) With Chemoradiation: Hispanic or Latino | 2
    Metformin (2000mg) With Chemoradiation: Not Hispanic or Latino | 4
    Metformin (2000mg) With Chemoradiation: Unknown or Not Reported | 0
    Metformin (2550mg) With Chemoradiation: number analyzed (Participants) | 8
    Metformin (2550mg) With Chemoradiation: Hispanic or Latino | 8
    Metformin (2550mg) With Chemoradiation: Not Hispanic or Latino | 0
    Metformin (2550mg) With Chemoradiation: Unknown or Not Reported | 0
    Metformin (3000mg) With Chemoradiation: number analyzed (Participants) | 4
    Metformin (3000mg) With Chemoradiation: Hispanic or Latino | 0
    Metformin (3000mg) With Chemoradiation: Not Hispanic or Latino | 4
    Metformin (3000mg) With Chemoradiation: Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: There is a total of 18 participants in three cohorts: Metformin (2000mg) (n = 6); Metformin (2500mg) (n = 8); Metformin (3000mg) (n = 4).
  Participants
    Metformin (2000mg) With Chemoradiation: number analyzed (Participants) | 6
    Metformin (2000mg) With Chemoradiation: American Indian or Alaska Native | 0
    Metformin (2000mg) With Chemoradiation: Asian | 0
    Metformin (2000mg) With Chemoradiation: Native Hawaiian or Other Pacific Islander | 0
    Metformin (2000mg) With Chemoradiation: Black or African American | 0
    Metformin (2000mg) With Chemoradiation: White | 6
    Metformin (2000mg) With Chemoradiation: More than one race | 0
    Metformin (2000mg) With Chemoradiation: Unknown or Not Reported | 0
    Metformin (2550mg) With Chemoradiation: number analyzed (Participants) | 8
    Metformin (2550mg) With Chemoradiation: American Indian or Alaska Native | 0
    Metformin (2550mg) With Chemoradiation: Asian | 0
    Metformin (2550mg) With Chemoradiation: Native Hawaiian or Other Pacific Islander | 0
    Metformin (2550mg) With Chemoradiation: Black or African American | 0
    Metformin (2550mg) With Chemoradiation: White | 8
    Metformin (2550mg) With Chemoradiation: More than one race | 0
    Metformin (2550mg) With Chemoradiation: Unknown or Not Reported | 0
    Metformin (3000mg) With Chemoradiation: number analyzed (Participants) | 4
    Metformin (3000mg) With Chemoradiation: American Indian or Alaska Native | 0
    Metformin (3000mg) With Chemoradiation: Asian | 0
    Metformin (3000mg) With Chemoradiation: Native Hawaiian or Other Pacific Islander | 0
    Metformin (3000mg) With Chemoradiation: Black or African American | 2
    Metformin (3000mg) With Chemoradiation: White | 2
    Metformin (3000mg) With Chemoradiation: More than one race | 0
    Metformin (3000mg) With Chemoradiation: Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 18
Tobacco Users [Count of Participants; unit: Participants] — Population: There is a total of 18 participants in three cohorts: Metformin (2000mg) (n = 6); Metformin (2500mg) (n = 8); Metformin (3000mg) (n = 4).
  Participants
    Metformin (2000mg) With Chemoradiation: number analyzed (Participants) | 6
    Metformin (2000mg) With Chemoradiation | 3
    Metformin (2550mg) With Chemoradiation: number analyzed (Participants) | 8
    Metformin (2550mg) With Chemoradiation | 7
    Metformin (3000mg) With Chemoradiation: number analyzed (Participants) | 4
    Metformin (3000mg) With Chemoradiation | 2

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of Metformin in Combination With Concurrent Cisplatin and Radiation
Description: Cohorts of patients received escalating doses of metformin (2000 mg, 2550 mg, or 3000 mg divided into daily doses) with a 7-day to 14-day lead-in prior to CRT based on the modified toxicity probability interval design to allow for possible re-escalation after previous de-escalation and to maximize the ability to identify the maximum tolerated dose (MTD). Patients continued to receive metformin for the duration of CRT as tolerated.
Time Frame: 24 months
Population: Proportion of the study sample that were evaulable.
Measure: Number; unit: mg
Groups:
- Metformin (2000mg) With Chemoradiation; Metformin (2550mg) With Chemoradiation; Metformin (3000mg) With Chemoradiation: Metformin administered orally daily to start one week prior to Cisplatin and Radiation Therapy. Metformin dose is escalating.
  Metformin: Escalating doses of 2000mg, 2550 mg and 3000mg. Starting 1 week prior to the initiation of chemoradiation and ending the final day of chemo or radiation.
  Cisplatin: Dosed at 100mg/m2 on days 1, 22, and 43
  Radiation Therapy: 70 Gy in 2 Gy once daily fractions of 35 fractions
Arm/Group | Metformin (2000mg) With Chemoradiation | Metformin (2550mg) With Chemoradiation | Metformin (3000mg) With Chemoradiation
Number analyzed (Participants) | 6 | 8 | 4
mg | NA — The MTD for metformin could not be established reliably from the current study. | NA — The MTD for metformin could not be established reliably from the current study. | NA — The MTD for metformin could not be established reliably from the current study.

2. Secondary Outcome: Number of Participants Experiencing No-Reoccurrence at 36 Months
Description: Patients were evaulated at 36 months to determine if there was recurrence of disease.
Time Frame: 36 months
Measure: Count of Participants; unit: Participants
Groups:
- Metformin (2000mg) With Chemoradiation: Metformin administered orally daily to start one week prior to Cisplatin and Radiation Therapy. Metformin dose is escalating. Metformin cohort: 2000mg.
- Metformin (2550mg) With Chemoradiation: Metformin administered orally daily to start one week prior to Cisplatin and Radiation Therapy. Metformin dose is escalating. Metformin cohort: 2550mg.
- Metformin (3000mg) With Chemoradiation: Metformin administered orally daily to start one week prior to Cisplatin and Radiation Therapy. Metformin dose is escalating. Metformin cohort: 3000mg.
Arm/Group | Metformin (2000mg) With Chemoradiation | Metformin (2550mg) With Chemoradiation | Metformin (3000mg) With Chemoradiation
Number analyzed (Participants) | 6 | 8 | 4
Participants | 6 | 8 | 4

3. Secondary Outcome: Number of Participants With Adverse Events
Description: Adverse event means any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. Adverse event means any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related.Any participants with any adverse event at any grade was included. Adverse events were collected during the on study period of 21 weeks up to three months after the study for a total of 34 weeks.
Time Frame: 36 months
Measure: Count of Participants; unit: Participants
Groups:
- Metformin (2000mg) With Chemoradiation: Subjects receiving Metformin (2000mg) along with chemoradiation.
- Metformin (2550mg) With Chemoradiation; Metformin (3000mg) With Chemoradiation: Subjects receiving Metformin (2500mg) along with chemoradiation.
Arm/Group | Metformin (2000mg) With Chemoradiation | Metformin (2550mg) With Chemoradiation | Metformin (3000mg) With Chemoradiation
Number analyzed (Participants) | 6 | 8 | 4
Participants | 6 | 7 | 4

4. Secondary Outcome: Progression Free Survival
Description: 2-year progression free survival
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Metformin (2000mg) With Chemoradiation | Metformin (2550mg) With Chemoradiation | Metformin (3000mg) With Chemoradiation
Number analyzed (Participants) | 6 | 8 | 4
Participants | 6 | 8 | 4

5. Secondary Outcome: Overall Survival
Description: 2 year overall survival
Time Frame: 24 months
Measure: Number; unit: participants
Arm/Group | Metformin (2000mg) With Chemoradiation | Metformin (2550mg) With Chemoradiation | Metformin (3000mg) With Chemoradiation
Number analyzed (Participants) | 6 | 8 | 4
participants | 5 | 8 | 4

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the on study period of 21 weeks up to three months after the study for a total of 34 weeks.
Groups:
- Metformin With Chemoradiation- 2000mg Cohort: Metformin administered orally daily to start one week prior to Cisplatin and Radiation Therapy. Metformin dose is escalating.
  Metformin: Escalating doses of 2000mg. Starting 1 week prior to the initiation of chemoradiation and ending the final day of chemo or radiation.
  Cisplatin: Dosed at 100mg/m2 on days 1, 22, and 43
  Radiation Therapy: 70 Gy in 2 Gy once daily fractions of 35 fractions
- Metformin With Chemoradiation- 2550mg Cohort: Metformin administered orally daily to start one week prior to Cisplatin and Radiation Therapy. Metformin dose is escalating.
  Metformin: Escalating doses of 2550 mg. Starting 1 week prior to the initiation of chemoradiation and ending the final day of chemo or radiation.
  Cisplatin: Dosed at 100mg/m2 on days 1, 22, and 43
  Radiation Therapy: 70 Gy in 2 Gy once daily fractions of 35 fractions
- Metformin With Chemoradiation- 3000mg Cohort: Metformin administered orally daily to start one week prior to Cisplatin and Radiation Therapy. Metformin dose is escalating.
  Metformin: Escalating doses of 3000 mg. Starting 1 week prior to the initiation of chemoradiation and ending the final day of chemo or radiation.
  Cisplatin: Dosed at 100mg/m2 on days 1, 22, and 43
  Radiation Therapy: 70 Gy in 2 Gy once daily fractions of 35 fractions
Arm/Group | Metformin With Chemoradiation- 2000mg Cohort | Metformin With Chemoradiation- 2550mg Cohort | Metformin With Chemoradiation- 3000mg Cohort
All-Cause Mortality (participants affected / at risk) | 1/6 | 0/8 | 0/4
Serious Adverse Events (participants affected / at risk) | 6/6 | 1/8 | 1/4
Other Adverse Events (participants affected / at risk) | 6/6 | 7/8 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metformin With Chemoradiation- 2000mg Cohort (N=6) | Metformin With Chemoradiation- 2550mg Cohort (N=8) | Metformin With Chemoradiation- 3000mg Cohort (N=4)
Lung infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Mucositis Oral (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Creatinine Increased (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metformin With Chemoradiation- 2000mg Cohort (N=6) | Metformin With Chemoradiation- 2550mg Cohort (N=8) | Metformin With Chemoradiation- 3000mg Cohort (N=4)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Acute Kidney Disease (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 4 (5) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0)
Alkaline phosphatase increased (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 3 (4) | 1 (1) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (3) | 0 (0) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 1 (1)
Creatinine increase (Hepatobiliary disorders) | 1 (3) | 0 (0) | 2 (2)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 3 (4)
Dry Mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dysgeusia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0)
Ear Pain (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Edema Trunk (General disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 2 (2) | 1 (1) | 3 (3)
Fever (General disorders) | 1 (1) | 0 (0) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Hearing impaired (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2) | 2 (3) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Thrush (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Throat Swelling (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)
Odynophagia (Investigations) | 2 (2) | 0 (0) | 1 (2)
Laryngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Lymphedema (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Lymphocyte count increased (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
VB12 deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 2 (3) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (4) | 4 (4) | 0 (0)
Nervous system disorders (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Paresthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Odgnophagia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (2)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (5) | 0 (0)
Stomach Pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 2 (2) | 4 (4) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 2 (2) | 3 (3)
Weight Loss (Investigations) | 0 (0) | 1 (1) | 0 (0)
White blood cell decreased (Investigations) | 3 (3) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-08-31): https://cdn.clinicaltrials.gov/large-docs/01/NCT02325401/Prot_SAP_000.pdf
  • Informed Consent Form (2018-02-07): https://cdn.clinicaltrials.gov/large-docs/01/NCT02325401/ICF_001.pdf